CLINICAL TRIAL: NCT04241055
Title: Can a Values Affirmation Improve the Classroom Outcomes and Well-being of K-12 Teachers?
Brief Title: Values Affirmation to Improve Teachers' Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic, the primary dependent variables could not be collected as designed in the research plan
Sponsor: Wake Forest University (Other)
Collaborators: Stanford University (Other); Relay Graduate School of Education (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: WakeFU
Record Dates: First submitted 2019-10-04; First posted 2020-01-27 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will not know what the conditions are or which they are in. Staff from the collaborating organization will not know which conditions participants are in, and most staff members will not know details of the study. Researchers will not know which condition participants are in if/when they interact with participants (e.g., through email).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The "control" condition of a standard values affirmation intervention
  Interventions: Behavioral: Active control exercise
- Values affirmation (Experimental): The "treatment" condition of a standard values affirmation intervention
  Interventions: Behavioral: Values affirmation exercise

INTERVENTIONS:
Behavioral: Values affirmation exercise — In the experimental values affirmation condition, participants spend 10-15 minutes completing a guided reflection regarding values that are personally important (see Logel and Cohen, 2012; Brady, Griffiths, & Cohen, in prep).
  Arms: Values affirmation
Behavioral: Active control exercise — In the active control condition, participants spend 10-15 minutes completing a guided reflection regarding values that are not personally important but could be important to someone else (see Logel and Cohen, 2012; Brady, Griffiths, & Cohen, in prep).
  Arms: Control

SUMMARY:
The purpose of this project is to examine whether a values affirmation intervention improves teacher-student relationships, classroom performance, and well-being of first-year teachers.

ELIGIBILITY:
Inclusion Criteria:

* Must be teachers (current or prospective) affiliated with the Relay Graduate School of Education in the targeted classes/programs
* Must consent to participate and begin the experimental (values affirmation or control) exercise

Exclusion Criteria:

* None

Note: Our primary hypotheses focus on the effects of values affirmation for first-year teachers, particularly White first-year teachers at majority minority schools. Participants who are not White first-year teachers will be permitted in the study, but will not be included in confirmatory analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Student-teacher relationships | Approximately 6 months post-intervention
  Teachers will complete a survey that includes a 4-item scale to assess the quality of their relationships with students (scale: 1=not at all true for me; 5=extremely true for me)
  1. I have a good relationship with my students.
  2. My students have a positive opinion of me.
  3. I feel comfortable interacting with my students.
  4. My students respect me.
Teacher well-being | Approximately 6 months post-intervention
  Teachers will complete a survey that assesses their well-being. Average scores for the individual scales (below) will be computed. Scales will then be averaged to create a composite score. Due to space constraints, the full text of the scales is available on the project's OSF page at https://osf.io/ju5gh/.
  Burnout (7 items; scale: 1=not at all true for/of me, 5=very much true for/of me; reverse-scored for composite)
  Self-integrity (3 items; scale: 1=strongly disagree, 7=strongly agree)
  Belonging (3 items; scale: 1=strongly disagree, 7=strongly agree)
  Belonging uncertainty (2 items; scale: 1=strongly disagree, 7=strongly agree) [reverse-scored for composite]
  Perceived stress (4 items; scale: 1=never, 5=very often) [reverse-scored for composite]
Classroom Assessment Scoring System (CLASS) - "Instructional Support" dimension | Approximately 6 months post-intervention
  To assess quality of teachers' instruction, we will use the "instructional support" dimension of the CLASS (https://curry.virginia.edu/classroom-assessment-scoring-system). Coding will be conducted by staff from the Relay Graduate School of Education or their designees.

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University (via online survey tool), Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided